CLINICAL TRIAL: NCT04488315
Title: Pre-emptive Scalp Infiltration With Dexamethasone Lipid Microsphere Plus Ropivacaine for Postoperative Pain After Craniotomy
Brief Title: Scalp Infiltration With Dexamethasone Plus Ropivacaine for Post-craniotomy Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Day Surgery and Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY-2018-034-02-8
Record Dates: First submitted 2020-07-19; First posted 2020-07-28 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The dexamethasone lipid microsphere plus ropivacaine group (Experimental)
  Interventions: Drug: Dexamethasone lipid microsphere plus ropivacaine
- The ropivacaine alone group (Active Comparator)
  Interventions: Drug: Ropivacaine alone

INTERVENTIONS:
Drug: Dexamethasone lipid microsphere plus ropivacaine — Local scalp infiltration solution will consist of 30ml miscible liquids containing 8 mg dexamethasone lipid microsphere, 150mg ropivacaine and normal saline.
  Other Names: ropivacaine plus D-PAL
  Arms: The dexamethasone lipid microsphere plus ropivacaine group
Drug: Ropivacaine alone — Local scalp infiltration solution will consist of 30ml miscible liquids containing 150mg ropivacaine and normal saline
  Arms: The ropivacaine alone group

SUMMARY:
According to recent studies, patients following craniotomy suffer more than minimal pain; two-thirds of patients experienced moderate to severe pain. Postoperative pain most often occurs within 48 hours after surgery. Local infiltration of anesthesia is the most simple and effective analgesia. However, the analgesic effect only lasts for a short-time after surgery, and it cannot adequately meet the needs of postoperative analgesia after craniotomy. Several studies have shown that the mixture of dexamethasone with local anesthetics could reduce the postoperative pain scores better than local anesthetics alone. Lipid microsphere is a relatively new drug delivery system. It is an artificial lipid emulsion. Studies have shown that dexamethasone lipid microsphere, the dexamethasone palmitate emulsion (D-PAL emulsion), has stronger anti-inflammatory effect than dexamethasone. Therefore, the investigators hypothesize that the pre-emptive scalp infiltration with dexamethasone lipid microsphere plus ropivacaine could achieve superior postoperative pain-relief compared to ropivacaine alone for patients undergoing craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective craniotomy under general anesthesia;
* Age 18-64 years;
* American Society of Anesthesiologists (ASA) physical status of I or II;
* Anticipated tracheal extubation, full recovery and cooperation within 2 hours postoperatively
* Patients required to fix their head in a head clamp during the operation.

Exclusion Criteria:

* Previous history of craniotomy;
* Plan to delay extubation or no plan to extubate;
* Patients who cannot use the patient-controlled analgesia (PCA) device;
* Patients who cannot comprehend the instructions of a numeric rating scale (NRS) before craniotomy;
* Body mass index (BMI) <15 or >35;
* Allergy to dexamethasone, lipid microsphere, opioids or ropivacaine;
* History of drug abuse or excessive alcohol, chronic opioids use (more than 2 weeks), or use of any sedative or analgesic before surgery;
* History of uncontrolled epilepsy, psychiatric disorders or chronic headache;
* Pregnant or at breastfeeding;
* Symptomatic cardiopulmonary, liver or renal dysfunction or combined with diabetes or other systemic dysfunction;
* Glasgow Coma Scale <15 before the surgery;
* Intracranial hypertension;
* Peri-incisional infection;
* Patients who have received chemoradiotherapy before the surgery or expected to receive postoperative chemoradiotherapy according to the preoperative imaging.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
The pain NRS scores at 24 h after craniotomy | At 24 hours after the operation
  The numeral rating scale allows a person to describe the intensity of the pain as a number usually ranging from 0 to 10, where "0" means "no pain" and "10" means pain as "bad as it could be".

SECONDARY OUTCOMES:
The first time the patients press the PCA button | Within 24, 48,72 hours postoperatively
  Patients will use PCA device for postoperative analgesia. When the patients feel pain, the PCA button will be pressed. The PCA device will provide a bolus of 2μg sufentanil with a 10 minutes lock-out time, and the maximum dose of sufentanil will be limited to 8μg/h.
The number of patients who didn't press the PCA button | Within 24, 48, 72 hours postoperatively
  Patients will use PCA device for postoperative analgesia. When the patients feel pain, the PCA button will be pressed. The PCA device will provide a bolus of 2μg sufentanil with a 10 minutes lock-out time, and the maximum dose of sufentanil will be limited to 8μg/h.
The number of times patients press the PCA button | Within 24, 48, 72 hours postoperatively
  Patients will use PCA device for postoperative analgesia. When the patients feel pain, the PCA button will be pressed. The PCA device will provide a bolus of 2μg sufentanil with a 10 minutes lock-out time, and the maximum dose of sufentanil will be limited to 8μg/h.
The NRS score | At 2 hours, 4 hours, 12 hours, 48 hours, 72 hours, 1 month, and 3 months after the operation
  The numeral rating scale allows a person to describe the intensity of the pain as a number usually ranging from 0 to 10, where "0" means "no pain" and "10" means pain as "bad as it could be".
The incidence of PONV | Within 24, 48, 72 hours after surgery
  Postoperative nausea and vomiting: 0 represents absent; 1 represents nausea without treatment; 2 represents nausea in need of treatment; 3 represents vomiting
Time to first rescue analgesia with OC/APAP after surgery | At 2 hours, 4 hours, 8 hours, 24 hours and 48 hours postoperatively
  Patients will be given an oral supplementary tablet of oxycodone (OC)/acetaminophen (APAP) 5/325-mg (MallinckrodtInc.USA) for rescue analgesia when NRS score > 4 after receiving four times of bolus with the PCA device. OC/ APAP will be prescribed at an interval of at least 6 h until the end of our study.
Duration of hospitalization | From the date of the surgery until the date of discharge, assesses up to 7 days
  From the date of the surgery until the date of discharge
WHOQOL-BREF scores | At 1 month and 3 months after surgery
  The World Health Organization QoL abbreviated version scale consists of 26 items and involves 4 aspects: A. Physical health (7 items); B. Psychological health (6 items); C. Social relationships (3 items); D. Environment (8 items). Other two items measure the patients' quality of life and general health. The average score for each domain can range from 4 to 20, and the higher the score, the better the quality of life.
Wound healing scores | At 1 and 3 months after surgery
  Wound healing scores： 1 represents skin fully healed, no infection, hair regrowth along wound; 2 represents skin ≤3cm in total not healed, ≤0.5cm margin of redness, hair ≤3cm not regrowthing; 3 represents skin >3cm not healed, more redness or superficial pus, >3-6cm not regrowthing hair; 4 represents areas of necrosis ≤3cm, deep infection, >6cm not regrowthing hair; 5 represents areas of necrosis >3cm.
POSAS scores | At 3 months after surgery
  The Patient and Observer Scar Assessment Scale consists of two scales: the observer scale and the patient scale. Both scales contain six items that are scored numerically. Each of the six items on both scales has a 10-step score, with 10 indicating the worst imaginable scar or sensation. The total score of both scales consists of adding the scores of each of the six items (range, 6 to 60). The lowest score, 6, reflects normal skin, whereas the highest score, 60, reflects the worst imaginable scar.
Adverse events | Through the whole follow-up, an average of 3 months
  Steroid-hormone related complications, such as wound infection, wound edema, delayed wound healing, pulmonary infections, gastric ulcers, local atrophy or infection, embolic events and so on
Cumulative sufentanil consumption by PCA device | During 24hours, 48 hours and 72 hours postoperatively
  A Patient Controlled Analgesia (PCA) device containing sufentanil 200μg and ondansetron 16 mg in 100 ml saline will be set up to deliver 1 mL as an intravenous bolus with a 10-min lockout interval after craniotomy. The maximum dose will be limited to 8 μg per hour, and there will be no initial dose or background infusion. Patients will be advised to push the analgesic demand button if they feel pain and to repeat it until the pain is relieved.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Principal Investigator — Beijing Tian Hospital; Wei Zhang, MD, Principal Investigator — Beijing Tian Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Zhou H, Ou M, Yang Y, Ruan Q, Pan Y, Li Y. Effect of skin infiltration with ropivacaine on postoperative pain in patients undergoing craniotomy. Springerplus. 2016 Jul 26;5(1):1180. doi: 10.1186/s40064-016-2856-3. eCollection 2016. PMID 27512639
- [Background] Gottschalk A, Berkow LC, Stevens RD, Mirski M, Thompson RE, White ED, Weingart JD, Long DM, Yaster M. Prospective evaluation of pain and analgesic use following major elective intracranial surgery. J Neurosurg. 2007 Feb;106(2):210-6. doi: 10.3171/jns.2007.106.2.210. PMID 17410701
- [Background] Jia Y, Zhao C, Ren H, Wang T, Luo F. Pre-emptive scalp infiltration with dexamethasone plus ropivacaine for postoperative pain after craniotomy: a protocol for a prospective, randomized controlled trial. J Pain Res. 2019 May 24;12:1709-1719. doi: 10.2147/JPR.S190679. eCollection 2019. PMID 31213883
- [Derived] Zhang W, Li C, Zhao C, Ji N, Luo F. Pre-incisional infiltration with ropivacaine plus dexamethasone palmitate emulsion for postoperative pain in patients undergoing craniotomy: study protocol for a prospective, randomized controlled trial. Trials. 2022 Dec 12;23(1):996. doi: 10.1186/s13063-022-06936-z. PMID 36510271